CLINICAL TRIAL: NCT06308926
Title: A Phase IIa, Double-Blind, Randomized, Multi-Center Study Comparing MRG-001 to Placebo in Patients With Acute Respiratory Distress Syndrome
Brief Title: MRG-001 as an Immunoregulatory and Regenerative Therapy for ARDS Patients
Acronym: SUMMIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedRegen LLC (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRG23ARDS
Record Dates: First submitted 2023-12-18; First posted 2024-03-13 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Distress Syndrome; Respiratory Failure; Respiratory Distress Syndrome; Respiratory Tract Diseases; Cytokine Storm
Keywords: Acute Respiratory Distress Syndrome; MRG-001; Stem Cells; Immunomodulation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Respiratory Tract Diseases; Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MRG-001 (Low-dose) (Experimental): MRG-001 will be administered subcutaneously at 0.007 mL/kg. Patients will receive 3 injections per week every other day for a total of 2 weeks or until discharge from the ICU.
  Interventions: Drug: MRG-001 (Low-dose)
- MRG-001 (High-dose) (Experimental): MRG-001 will be administered subcutaneously at 0.01 mL/kg. Patients will receive 3 injections per week every other day for a total of 2 weeks or until discharge from the ICU.
  Interventions: Drug: MRG-001 (High-dose)
- Placebo (Placebo Comparator): Sterile injectable saline will be administered subcutaneously at 0.01 mL/kg. Patients will receive 3 injections per week every other day for a total of 2 weeks or until discharge from the ICU.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MRG-001 (Low-dose) — MRG-001 is subcutaneously administered.
  Arms: MRG-001 (Low-dose)
Drug: MRG-001 (High-dose) — MRG-001 is subcutaneously administered.
  Arms: MRG-001 (High-dose)
Other: Placebo — Saline placebo will be administered subcutaneously based on bodyweight and similar dose as the treatment group.
  Arms: Placebo

SUMMARY:
This is a phase IIa, dose-ranging, proof-of-concept study of MRG-001 in patients with ARDS.

The aim is to determine the safety and preliminary efficacy of MRG-001 across two dose ranges.

ELIGIBILITY:
Inclusion Criteria:

Acute Respiratory Distress Syndrome, manifested by the following and not explained by alternative diagnoses, for example but not limited to: Pulmonary Edema due to Congestive Heart Failure (CHF).

1. Chest x-ray (CXR)* revealing bilateral infiltrates involving a minimum of three quadrants on frontal chest radiograph, consistent with pulmonary edema or bilateral ground glass opacities not fully explained by effusions, lobar or lung collapse, nodules, atelectasis or other etiology of infiltrates not due to ARDS.
2. PaO2/FiO2 < 300.
3. Requiring respiratory support [defined as mechanical ventilation, non-invasive ventilation (NIV) or high flow nasal canula (HFNC)] If on ventilator, settings must include positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP) ≥5 cm H2O.

Exclusion Criteria:

1. Age less than 18 years.
2. Infiltrates with etiology suspected of mimicking ARDS, ie; Pulmonary Edema due to Congestive Heart Failure (CHF). (A Pulmonary Arterial Wedge Pressure (PAWP) of < 18 for >12 hours would rule out suspected CHF).
3. Pregnancy documented or suspected in women of child bearing potential, unless ruled out by a negative pregnancy test during screening or breast feeding.
4. Immunocompromised patients:

   4.1. Organ or bone marrow transplant recipients and/or recent (within 2 months) chronic use of immunosuppressive drugs (tacrolimus, mycofenolate mofetil, cyclosporine, rapamycine, hydrochloroquine, azathiopurine, methotrexate), e.g., biologicals, JAK1/2 inhibitors, interferons, interleukins, (prednisone or related corticosteroids are allowed).

   4.2. Patients with documented or suspected HIV/AIDS, hepatitis B/C or active lung disease with tuberculosis. 4.3. Patients with active cancer diagnosis or use of chemotherapy in the past 3 months.
5. Hypersensitivity to either of the components of MRG-001.
6. The patient is known or suspected to be brain dead or is moribund (not expected to live >48 hours) or is unlikely to survive long enough to receive 3 injections (4 days) in the opinion of the investigator.
7. The primary care physician is not committed to full support of the patient. (A DNR representing "no chest compression" only, would not necessarily be an exclusion. A DNR in which life support is withheld/withdrawn or is otherwise limited, would be an exclusion).
8. Participation in another investigational protocol or use of another investigational drug within 30 days of enrollment.
9. Enrollment time window has been exceeded (must be enrolled within 7 days of hospital admission and within 48 hours of development of ARDS).
10. Significant pre-existing organ dysfunction prior to randomization:

    10.1. Lung: Receiving supplemental home oxygen therapy at baseline for pre-existing medical condition (other than COVID-19), as documented in medical record. 10.2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record. Clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction (past 3 months), heart and coronary vessel surgery (past 3 months), significant valvular heart disease, uncontrolled arterial hypertension with systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg. WHO Class III or IV pulmonary hypertension. 10.3. Renal: End-stage renal disease requiring renal replacement therapy or eGFR <30 mL/min. 10.4. Liver: Severe chronic liver disease defined as Child-Pugh Class C or pre-existing severe hepatic dysfunction (i.e.; portal hypertension, cirrhosis, ascites, esophageal variceal bleeding, acute hepatic necrosis). 10.5. Hematologic: Baseline platelet count <30,000/mm3 or hemoglobin levels <6.0 g/dL. 10.6. Neurological: Severe traumatic brain injury, with intracranial injury demonstrated by head CT 10.7. History of splenectomy or splenomegaly (spleen weighing > 750 g).
11. Currently receiving extracorporeal life support (ECLS/ECMO) or high-frequency oscillatory ventilation (HFOV).
12. Anticipated extubation within 24 hours of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Hemopoietic stem cell mobilization | 24 Hours
  The primary efficacy endpoint is the absolute change of hematopoietic stem cell mobilization (CD34+ cells) calculated as cells/μl at the peak of mobilization at 12 hours compared to baseline after MRG-001 injection. degree of hematopoietic stem cell mobilization (CD34+, cells/μl) measured as a longitudinal outcome over the first 24 hours after after MRG-001 injection.
Organ Failure | 28 Days
  The primary safety endpoint is organ system failure free days to day 28. Patients will be monitored daily for 28 days for signs of the failure of non-pulmonary organs and systems. The following non-pulmonary organ system failures will be assessed: circulatory, coagulation, hepatic and renal failure.

SECONDARY OUTCOMES:
Pharmacokinetics | 28 Days
  Change in the trough concentration (Ctrough) of tacrolimus in ng/mL in whole blood during the course of treatment.
Pharmacokinetics | 28 Days
  Change in the trough concentration (Ctrough) of plerixafor in ng/mL in plasma during the course of treatment.
Pharmacodynamics | 28 Days
  Change in absolute numbers or percentages from baseline in circulating stem cells and immune cells measured by flow cytometry
Cytokine Changes | 28 Days
  Change from baseline in serum cytokines including IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-17, IL-18, IFN- γ, TNF-α.
Respiratory-Free Days | 28 Days
  The number of days patients in the ICU do not require supplemental forms of oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon R Bernard, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmadi AR, Atiee G, Chapman B, Reynolds L, Sun J, Cameron AM, Wesson RN, Burdick JF, Sun Z. A phase I, first-in-human study to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of MRG-001 in healthy subjects. Cell Rep Med. 2023 Sep 19;4(9):101169. doi: 10.1016/j.xcrm.2023.101169. Epub 2023 Aug 25. PMID 37633275